CLINICAL TRIAL: NCT05020184
Title: Effect of Oral Cimetidine in the Protoporphyrias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amy K. Dickey, M.D. (Other)
Collaborators: Wake Forest University Health Sciences (Other); The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor-Investigator, Amy K. Dickey, M.D., Instructor of Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P002095; PC7211 (Other: Porphyrias Consortium Protocol Number); 1R01FD007287-01 (FDA)
Record Dates: First submitted 2021-07-26; First posted 2021-08-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Erythropoietic Protoporphyria; X-linked Protoporphyria
Keywords: Erythropoietic Protoporphyria; X-linked Protoporphyria; EPP; Cimetidine; Photosensitivity
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Protoporphyria, Erythropoietic, X-Linked Dominant; Photosensitivity Disorders | interventions — Cimetidine

STUDY DESIGN:
Intervention Model Description: The study design is a multicenter, prospective, randomized, double-blind, placebo-controlled, crossover trial of oral cimetidine 800mg twice daily versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cimetidine (Active Comparator): Cimetidine 800mg orally twice daily
  Interventions: Drug: Cimetidine
- Placebo (Placebo Comparator): Placebo capsule orally twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cimetidine — Oral Cimetidine 800mg twice daily.
  Other Names: Tagament
  Arms: Cimetidine
Drug: Placebo — Placebo twice daily
  Arms: Placebo

SUMMARY:
Erythropoietic protoporphyria (EPP) and X-linked protoporphyria (XLP) result from genetic defects of heme biosynthesis that cause life-long, painful cutaneous sensitivity to light. The objective of this study is to determine the efficacy and safety of oral cimetidine administration for treatment of the protoporphyrias. Efficacy will be based on protoporphyrin levels, photosensitivity, and quality of life questionnaires.

Funding Source- FDA OOPD

DETAILED DESCRIPTION:
Erythropoietic protoporphyria (EPP) and X-linked protoporphyria (XLP) are genetic defects of heme biosynthesis that cause life-long, painful cutaneous sensitivity to light. EPP and XLP, collectively called the protoporphyrias, result in the accumulation of the light-sensitive molecule protoporphyrin IX initially in the bone marrow during hemoglobin synthesis and secondarily in erythrocytes, plasma, and the liver. In addition to photosensitivity, protoporphyria can also result in anemia, gallstones, and liver failure. No therapy has been demonstrated to reduce protoporphyrin levels or prevent the potentially life-threatening complications of EPP. Cimetidine has gained attention as a possible treatment for human porphyrias because of a potential off-target effect of inhibition of delta-aminolevulinate synthase (ALAS), the first enzyme of heme biosynthesis. This inhibition was first described in vitro; however, case reports of benefit in EPP have been anecdotal and uncontrolled. Therefore, the objective of this study is to determine the efficacy and safety of oral cimetidine administration in the protoporphyrias. Efficacy will be based on protoporphyrin levels, photosensitivity, and quality of life questionnaires. If the results are positive, this would be the first study providing quality evidence for an agent acting as a disease-modifying therapy for EPP. The study is also attractive because it repurposes an already approved drug with few side effects to treat a rare human disease.

The study design is a prospective, blinded, randomized, 2x2 cross-over design comparing cimetidine to placebo in patients with protoporphyria. Eligible protoporphyria patients will be randomized with equal allocation to one of two treatment sequences that will be administered over two 3-month study periods. Randomization will be stratified by site and permuted block randomization will be used to prevent chronological bias. Patients randomized to sequence 1 will receive placebo during period 1 and cimetidine during period 2. Patients randomized to sequence 2 will receive cimetidine during period 1 and placebo during period 2. Between periods, to eliminate any carry-over effects from the treatment administered in period 1, a wash-out period of 3 months will occur in which all patients receive neither cimetidine nor placebo. Three months was selected for each study period and for the wash-out period because of the rapid decline in protoporphyrin in red cells over the lifespan of the red cell (120 days), as well as to account for the time frame needed to measure light sensitivity in EPP.

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment or co-enrollment in the Longitudinal Study of the Porphyrias (PC Study 7201) with a confirmed diagnosis of EPP or XLP
* Male or female age ≥15 years at screening
* Characteristic history of non-blistering cutaneous photosensitivity
* Willing and capable of giving informed consent and following procedures described in the protocol

Exclusion Criteria:

* Participants not willing to expose themselves to light to the point of prodromal symptoms at least weekly
* History of liver or bone marrow transplant or clinically significant liver dysfunction as determined by the Investigator
* Known or suspected allergy or intolerance to cimetidine
* Use of any other experimental therapy in the past 3 months at screening
* Use of cimetidine within the past 3 months at screening
* Individuals with elevations of porphyrins in plasma or erythrocytes due to other diseases (i.e., secondary porphyrinemia) such as liver and bone marrow diseases
* Patients with any clinically significant comorbid conditions, which in the opinion of the Investigator, precludes participation
* Treatment with any drugs or supplements (Appendix 1) that in the opinion of the Investigator can interfere with subject safety or the objectives of the study
* The participant either does not have a smartphone or is not willing to use his/her smartphone for the study
* Women who are pregnant, breastfeeding, or actively planning to become pregnant
* Individuals with moderate to severe renal insufficiency

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Erythrocyte total protoporphyrin level | Before and after each 3-month treatment period
  Percent change in erythrocyte total protoporphyrin level post-treatment relative to pre-treatment

SECONDARY OUTCOMES:
Time to prodrome | Last 2 months of each treatment period
  Time to prodrome measured as prodrome-free outdoor exposure time
Patient-reported quality of life | Before and after each 3-month treatment period
  Patient-reported quality of life as measured by Patient-Reported Outcomes Measurement Information System-57 (PROMIS-57) scale [0-100, where 100 is the best quality of life]
Phototoxic episodes | Last 2 months of each treatment period
  The number and severity of sunlight-induced pain events (phototoxic episodes)
Light dose | Last 2 months of each treatment period
  Light dose required for time to prodrome

CONTACTS AND LOCATIONS:
Overall Officials: Amy K Dickey, MD, Principal Investigator — Massachusetts General Hospital; Karl Anderson, MD, Principal Investigator — University of Texas
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, as well as the study protocol and statistical analysis plan, may be shared, after de-identification (text, tables, figures, and appendices), if meeting the time frame and access criteria listed below.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: With whom: Researchers who provide a methodologically sound proposal that is approved by the study investigators For what type of analysis: To achieve the aims of the approved proposal. By what mechanisms will the data be available: Proposals should be directed to adickey@mgh.harvard.edu . To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (3):
  • Informed Consent Form: Wake Forest Consent (2025-03-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT05020184/ICF_000.pdf
  • Informed Consent Form: UTMB Consent Form (2025-03-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT05020184/ICF_001.pdf
  • Informed Consent Form: MGH Consent form (2025-03-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT05020184/ICF_002.pdf